CLINICAL TRIAL: NCT01192997
Title: A Phase 2/3, Open Label, Randomised Study of the Safety, Reactogenicity and Immunogenicity of a Single Dose of Novartis Meningococcal ACWY (Menveo) or GSK Meningococcal ACWY Conjugate Vaccine in Adolescents Primed With Meningitec, Menjugate or Neisvac-C in Preschool Vaccination
Brief Title: Comparison of Two Meningococcal ACWY Conjugate Vaccines
Acronym: PRIME
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRIME
Record Dates: First submitted 2010-08-31; First posted 2010-09-01 (Estimated); Last update posted 2020-10-01 (Actual); Status verified 2018-08

CONDITIONS: Meningococcal Meningitis
Keywords: Meningitis; Meningococci; Meningitis C; Meningitis A; Meningitis W135; Meningitis Y; Antibody
MeSH Terms: conditions — Meningitis, Meningococcal; Meningitis | interventions — Meningococcal Vaccines; tetravalent meningococcal serogroups A, C, W-135 and Y tetanus toxoid conjugate vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Menveo-Meningitec (Active Comparator): Subjects who were primed with Meningitec who will receive Novartis Menveo
  Interventions: Biological: Menveo
- MenACWY-TT-Meningitec (Active Comparator): Subjects who were primed with Meningitec who will receive GSK MenACWY-TT
  Interventions: Biological: MenACWY-TT
- Menveo-Menjugate (Active Comparator): Subjects who were primed with Menjugate who will receive Novartis Menveo
  Interventions: Biological: Menveo
- MenACWY-TT-Menjugate (Active Comparator): Subjects who were primed with Menjugate who will receive GSK MenACWY-TT vaccine.
  Interventions: Biological: MenACWY-TT
- Menveo-NeisVac-C (Active Comparator): Subjects who were primed with NeisVac-C who will receive Novartis Menveo
  Interventions: Biological: Menveo
- MenACWY-TT-NeisVac-C (Active Comparator): Subjects who were primed with NeisVac-C who will receive GSK MenACWY-TT vaccine
  Interventions: Biological: MenACWY-TT

INTERVENTIONS:
Biological: Menveo — Single dose Menveo (a MenACWY vaccine conjugated to CRM-197).
  Arms: Menveo-Meningitec; Menveo-Menjugate; Menveo-NeisVac-C
Biological: MenACWY-TT — Single dose MenACWY-TT (MenACWY vaccine conjugated to Tetanus Toxoid, TT)
  Arms: MenACWY-TT-Meningitec; MenACWY-TT-Menjugate; MenACWY-TT-NeisVac-C

SUMMARY:
There is evidence of waning immunity in individuals vaccinated against meningitis C as part of the UK infant immunisation schedule. The intention of this study is to contact participants of a previous NVEC (National Vaccine Evalutaion Consortium) clinical trial (a PreSchool Men C trial, in which participants were randomised to receive Meningitec, Menjugate or Neisvac-C). They will be invited to enrol and will be randomised to receive one of two quadrivalent meningococcal ACWY vaccines, to look at the boosting effect they may confer.

DETAILED DESCRIPTION:
Between 550 and 650 subjects enrolled in a previous Meningococcal C vaccine study will be invited to join this new study looking at the boosting effects of two quadrivalent meningococcal ACWY vaccines. If they choose to participate, they will be randomised to receive one of the ACWY vaccines. Within each vaccine group, there will be further division into short (6 months) or longer (9 months) follow-up.

Each participant will be given one dose of an allocated vaccine. Blood samples will be taken three times from each participant - the first sample will be pre-vaccination; the second sample will be taken one month after vaccination; and the third and final sample at either six or nine months after vaccination (depending on the group they are randomised to).

ELIGIBILITY:
Inclusion Criteria:

* Previously enrolled on the Preschool Men C study conducted by NVEC in 1999/2000
* Participant's parent or legally authorized representative is willing and able to give written informed consent for participation after the nature of the study has been explained.
* No contraindications to vaccination as specified in the "Green Book"- Immunisation against Infectious Disease, HMSO.
* Participant who gives assent for participation in the study.
* Vaccinated with Meningitec (MCC CRM) or Menjugate (MCC CRM) or NeisVac-C (MCC TT) between 3.5-6 years of age.
* Known to be free of medical problems as determined by a medical history and clinical assessment.
* Parent or legally authorised representative is willing to allow his or her child's GP to be notified of participation in the study and contacted if required for confirmation of vaccination history.

Exclusion Criteria:

* History of invasive meningococcal disease.
* Have a history of household contact or intimate exposure to an individual with culture proven Neisseria meningitis disease in the previous 60 days.
* Any vaccination against MenC disease since MCC vaccine given between 3.5 to 6 years.
* Participant is pregnant.
* Confirmed or suspected immunosuppressive or immunodeficient conditions, including human immunodeficiency virus (HIV) infection.
* Major congenital defects or serious chronic disease including progressive neurological disease or seizure disorder.
* Have a known bleeding diathesis, or any condition that may be associated with a prolonged bleeding time.
* Have a history of severe allergic reactions after previous vaccinations such as anaphylactic shock, asthma, urticaria, or other allergic reaction or hypersensitivity to any vaccine component.
* Have received another investigational agent within 90 days or before completion of the safety follow-up period in another study, whichever is longer, prior to enrollment and unwilling to refuse participation in another investigational trial through the end of the study.
* In the event that administration of another licensed vaccine is needed during the study, this vaccine should not be administered within 30 days of any study injection according to investigator's judgment (exception: licensed flu-vaccine should not be administered within 14 days of study vaccines).
* Have received any blood or blood products within the past 12 weeks.
* Have any other significant disease or disorder which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Temporary Exclusion Criteria

• Receipt of systemic antibiotics (either oral or parenteral) will delay enrolment until at least 7 days after cessation of antibiotics.

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 91 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Response to meningococcal components of the vaccines by serum bactericidal antibody | December 2013
  Percentage of participants with serogroup-specific rabbit Serum Bactericidal Antibody (rSBA) titres ≥ 8 at one month post vaccination, for each of the serogroups A, C, W135 and Y. (This titre of rSBA is a documented correlate of protection for meningococcal conjugate vaccines)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MD, Study Chair — Public Health England
Locations (3):
- United Kingdom (3):
  - Multiple General Practice surgeries, Gloucester, Gloucestershire
  - Multiple General Practice surgeries, Hertford, Hertfordshire
  - Health Protection Agency, Immunisation Department, Colindale, London

REFERENCES:
- [Result] Ishola DA, Andrews N, Waight P, Yung CF, Southern J, Bai X, Findlow H, Matheson M, England A, Hallis B, Findlow J, Borrow R, Miller E. Randomized Trial to Compare the Immunogenicity and Safety of a CRM or TT Conjugated Quadrivalent Meningococcal Vaccine in Teenagers who Received a CRM or TT Conjugated Serogroup C Vaccine at Preschool Age. Pediatr Infect Dis J. 2015 Aug;34(8):865-74. doi: 10.1097/INF.0000000000000750. PMID 26075813
- See also: Published study results — http://www.ncbi.nlm.nih.gov/pubmed/26075813